CLINICAL TRIAL: NCT04329910
Title: Dynamic Surgical Conditions and Body Habitus Independently Impair Pulmonary Mechanics During Robotic Assisted Laparoscopic Surgery: A Cross-Sectional Study
Brief Title: Obesity Alters Lung Mechanics in Robotic Surgery
Status: Completed | Type: Observational
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, William G Tharp, Assistant Professor, University of Vermont Medical Center
Other Study IDs: M18-0048
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Surgery; Anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Lean: BMI < 25
  Interventions: Other: no intervention
- overweight: BMI 25 - 29.9
  Interventions: Other: no intervention
- class i obesity: BMI 30 -34.9
  Interventions: Other: no intervention
- class ii obesity: BMI 35 - 39.9
  Interventions: Other: no intervention
- class iii obesity: BMI >= 40
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention - observational only

SUMMARY:
Intraoperative lung protective ventilation strategies using standardized tidal volumes based on predicted body weight have proven beneficial, but attempts to standardize positive end expiratory pressure (PEEP) settings have not robustly accounted for body habitus or dynamic surgical conditions. Laparoscopic abdominal surgery in Trendelenburg (head-down) is an increasingly common surgical modality that presents a unique physiological challenge to the pulmonary system. In order to delineate the impact of body habitus, pneumoperitoneum, and surgical positioning on intraoperative pulmonary mechanics we conducted an observational study of patients undergoing robotic assisted laparoscopic abdominal surgery in Trendelenburg position. Using esophageal manometry, we partitioned the mechanical properties of the respiratory system into its lung and chest wall components and evaluated the effects of pneumoperitoneum, surgical position, and body mass index (BMI) on transpulmonary pressures, airway and transpulmonary driving pressures, and lung elastance. We hypothesized that increasing BMI would be associated with evidence of increasing atelectasis, increased driving pressures, and elevated lung elastance and that these changes would be exacerbated by pneumoperitoneum and Trendelenburg positioning.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were presentation for robotic assisted laparoscopic abdominal surgery in the supine position, age ≥ 18 years, and ability to provide informed consent

Exclusion Criteria:

* Exclusion criteria included intrinsic lung disease, ≥ 20 pack year smoking history, reactive airways disease, home oxygen requirement, inability to provide informed consent, emergent surgery, or esophageal pathology (i.e., strictures, varices, history of esophageal dilatation or surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robotic assisted laparoscopic abdominal surgery at the University of Vermont Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure | during the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vemont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No